CLINICAL TRIAL: NCT05248984
Title: Dosing of Ketorolac Impacts Post-cesarean paiN manaGemenet (KING): A Randomized Controlled Trial
Brief Title: Dosing of Ketorolac Impacts Post-cesarean paiN manaGemenet (KING)
Acronym: KING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kara M Rood, MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022H0063
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Post Cesarean Pain
Keywords: Postoperative pain; Cesarean; Ketorolac
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketorolac 30 mg (Active Comparator): Participants will receive single dose of intravenous (IV) Ketorolac 30mg
  Interventions: Drug: Ketorolac
- Ketorolac 60 mg (Active Comparator): Participants will receive single dose of intravenous (IV) Ketorolac 60mg
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Once the decision has been made by the primary obstetrics (OB) provider to proceed with cesarean delivery, participants will be randomized in to one of two groups:
  * Single dose of intravenous (IV) Ketorolac 30mg Vs.
  * Single dose of intravenous (IV) Ketorolac 60mg

SUMMARY:
This is a randomized controlled single blinded trial to compare the morphine milligram equivalents (MME) use in the first 24 hours postoperatively after cesarean section in patients receiving a single dose of 30 mg intravenous ketorolac vs. 60 mg intravenous ketorolac in the operating room after the end of surgery.

DETAILED DESCRIPTION:
Administration of a dose of ketorolac for postoperative pain management at end of cesarean is routine practice at our institution.

This is a randomized controlled single blinded trial at The Ohio State University comparing a single dose of 30 mg intravenous ketorolac vs. 60 mg intravenous ketorolac in the operating room immediately after cesarean section.

Potential study participants will be identified at the time of admission to Labor and Delivery unit. Inclusion criteria must be met, namely patient's age, mode of delivery via cesarean section. The decision for mode of delivery will be at the discretion of the primary obstetrics (OB) provider. Indications for cesarean delivery would be: scheduled cesarean due to history of previous uterine surgery including prior cesarean section, failed induction of labor, arrest of second stage of labor, non-reassuring fetal status.

Patients will be approached for consent and enrollment when decision is made to proceed for cesarean section by their primary provider. Patients with allergy to Non-steroidal anti-inflammatory drugs (NSAIDs), history of opioid use disorder, chronic pain disorders, or undergoing an emergent Cesarean section, will be excluded from the study.

Once the decision has been made by the primary obstetrics (OB) provider to proceed with cesarean delivery, participants will be randomized in to one of two groups:

* Single dose of IV Ketorolac 30mg Vs.
* Single dose of IV Ketorolac 60mg

The intervention and primary outcome will take place over the span of 24 hour post-cesarean. Once enrolled and randomized, patients will be given either 60 mg or 30 mg of IV ketorolac at the end of the procedure. All other obstetric care will be at the discretion of the primary provider, including but not limited to pain management postoperatively. Analysis will be by intent to treat. The secondary outcomes will be collected during the hospital stay until discharge.

ELIGIBILITY:
1. Inclusion criteria:

   * Pregnant individuals aged 18-45 with a viable single or twin intrauterine pregnancy
   * Cesarean section as the delivery mode
   * Regional anesthesia (Spinal, Epidural, Combined Spinal Epidural)
2. Exclusion criteria:

   * Known allergy or adverse reaction to Non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, or ketorolac
   * Patients with peptic ulcer disease, preexisting kidney or liver disease
   * Hemodynamically unstable due to hemorrhage
   * Acute or chronic pain disorder
   * Physician/provider or patient refusal
   * Estimated blood loss > 2000 mL
   * General anesthesia
   * Opioid use disorder
   * Emergent Cesarean delivery
   * Coagulation disorders
   * Active asthma
   * Patients weighing <50 kg

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Comparing the morphine milligram equivalents (MME) use in the first 24 hours. postoperatively after cesarean section | After cesarean surgery up to 24 hours.
  Comparing the morphine milligram equivalents (MME) use in the first 24 hours postoperatively after cesarean section in patients receiving a single dose of 30 mg intravenous ketorolac vs. 60 mg intravenous ketorolac in the operating room after the end of surgery.

SECONDARY OUTCOMES:
Comparing the morphine milligram equivalents (MME) use during hospital stay. | After cesarean surgery during hospital stay up to 2-3 days.
  Comparing the morphine milligram equivalents (MME) use during hospital stay postoperatively after cesarean section in patients receiving a single dose of 30 mg intravenous ketorolac vs. 60 mg intravenous ketorolac in the operating room after the end of surgery.
Comparing patient reported pain score assessment. | After cesarean surgery up to 24 hours.
  Comparing patient reported pain score assessment on a scale of 0-10 in the first 24 hours postoperatively after cesarean section in patients receiving a single dose of 30 mg intravenous ketorolac vs. 60 mg intravenous ketorolac in the operating room after the end of surgery.
Comparing the time to first administration of opioid pain medication postoperatively. | After cesarean surgery up to 2-3 days.
  Comparing the time to first administration of opioid pain medication postoperatively after cesarean section in patients receiving a single dose of 30 mg intravenous ketorolac vs. 60 mg intravenous ketorolac in the operating room after the end of surgery.
Evaluating adverse maternal outcomes. | After cesarean surgery during hospital stay up to 2-3 days.
  Evaluating adverse maternal outcomes (acute kidney injury, admission to intensive care unit, maternal death).
Evaluating type of skin incision. | After cesarean surgery during hospital stay up to 2-3 days.
  Evaluating type of skin incision (Pfannenstiel vs. Vertical Midline).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No